CLINICAL TRIAL: NCT04419064
Title: Confirmation of Ventilation and Intubation by Determination With Ultrasonography: A Multicenter Observational Study
Brief Title: Confirmation of Ventilation and Intubation by Determination With Ultrasonography
Acronym: COVID-US
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Kadlec Regional Medical Center (Unknown); The Cleveland Clinic (Other); Baylor College of Medicine (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Mourad Senussi, Clinical Instructor of Medicine, University of Pittsburgh
Other Study IDs: STUDY20050011
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Mechanical Ventilation
Keywords: intubation; bedside ultrasound; point-of-care ultrasound
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — Tracheal and lung ultrasonography

SUMMARY:
Chest radiography is the gold standard for confirming tracheal intubation. Bedside ultrasound can be a useful alternative. The investigators are conducting a multi-center, observational study from January 2019 to May 2020 (COVID-US Study) to determine the feasibility of tracheal and lung ultrasound in confirming endotracheal tube placement in the critically ill.

DETAILED DESCRIPTION:
Endotracheal intubation is an important aspect of managing critically ill patients. Chest radiography remains the gold standard for confirming endotracheal tube positioning, however, ultrasonography can be a useful alternative. The objective of this study is to determine the feasibility of a combination of tracheal and thoracic ultrasonography to confirm adequate positioning of endotracheal tube placement in a cohort of critically ill participants including those with novel coronavirus-2019.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> or equal to 18 years of age) requiring intubation and mechanical ventilation as a part of their routine care

Exclusion Criteria:

* Recent neck or chest surgery
* Cervical spine immobilization
* Lack of availability of operators or equipment for performing the ultrasound protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, > 18 years of age, undergoing intubation and mechanical ventilation from 4 multiple intensive care units from 4 different academic and community hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Concordance with next occurring chest radiograph | within 24 hours
  Adequate endotracheal tube position in agreement with chest radiograph

SECONDARY OUTCOMES:
Esophageal Intubation detection | within intubation attempt
  Number of esophageal intubations detected during intubation attempt
Right main or endobronchial intubation | within intubation attempt
  Number of right main stem intubations detected with ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Mourad H Senussi, MD, MS, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Kadlec Regional Medical Center, Richland, Washington

IPD SHARING:
Plan to Share IPD: No